CLINICAL TRIAL: NCT05239975
Title: A Randomized, Double-blind Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of SCTV01C (A Bivalent SARS-CoV-2 Trimeric Spike Protein Vaccine) in Population Aged ≥12 Years and Previously Vaccinated With Inactivated COVID-19 Vaccine
Brief Title: A Study of the Immunogenicity and Safety of SCTV01C in Population Aged ≥12 Years and Previously Vaccinated With Inactivated COVID-19 Vaccine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There was not a need to carry out a study in LAO any more.
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCTV01C-01-In-LAO-1
Record Dates: First submitted 2022-02-14; First posted 2022-02-15 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; SARS-CoV2 Infection
Keywords: COVID-19; SARS-CoV-2 infection; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTV01C (Experimental): Participants will be administrated one dose of SCTV01C on Day 0 and Day 180
  Interventions: Biological: SCTV01C
- Comirnaty (Active Comparator): Participants will be administrated one dose of Comirnaty on Day 0 and Day 180
  Interventions: Biological: Comirnaty

INTERVENTIONS:
Biological: SCTV01C — intramuscular injection
  Arms: SCTV01C
Biological: Comirnaty — intramuscular injection
  Arms: Comirnaty

SUMMARY:
The objective of this study is to evaluate the immunogenicity and safety of SCTV01C in participants aged ≥12 years and previously fully immunized with inactivated COVID-19 vaccine.

DETAILED DESCRIPTION:
This is a randomized, double-blind, approved vaccine-controlled Phase II booster study to evaluate the immunogenicity and safety of SCTV01C compared with Comirnaty in participants aged ≥12 years and previously fully immunized with inactivated COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥12 years old when signing ICF;
2. Participants who were fully vaccinated (2 doses) with inactivated COVID-19 vaccine (Sinopharm COVID-19 vaccine) and the interval between the last dose and this study vaccination is ≥3 months and ≤12 months;
3. The Participant and/or his legal guardian and/or his entrusted person can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. The subject and/or his legal guardian and/or his entrusted person have the ability to read, understand, and fill in record cards;
5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
6. Fertile men and women of childbearing age voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the study vaccination; the pregnancy test results of women of childbearing age are negative on screening.

Exclusion Criteria:

1. Previously diagnosed with COVID-19.
2. Presence of fever within 3 days before the study vaccination;
3. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or corresponding immunosuppressants;
4. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
5. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
6. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
7. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the first six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
8. Patients on antituberculosis therapy;
9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (except for skin basal cell carcinoma and carcinoma in-situ of cervix), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
11. Participants who received any immunoglobulin or blood products in the previous 3 months, or plan to receive similar products during the study;
12. Participants who received other investigational drugs within 1 month before the study vaccination;
13. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
14. Participants received other drugs used for prevention of COVID-19 (exception for Sinopharm COVID-19 vaccine) ;
15. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
16. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
17. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
18. Those who plan to donate ovum or sperms during the study period;
19. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
20. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
21. Those who are tested positive for HIV in terms of serology.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
GMT of neutralizing antibodies to Delta (B.1.617.2) variant on D28. | Day 28 after the study vaccination

SECONDARY OUTCOMES:
Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subpopulations on D28. | Day 28 after the study vaccination
Seroresponse rates of neutralizing antibodies of Delta (B.1.617.2) variant on D28. | Day 28 after the study vaccination
Seroresponse rates of neutralizing antibodies of Omicron (B.1.1.529) on D28. | Day 28 after the study vaccination
GMT of neutralizing antibodies to Omicron (B.1.1.529) variant on D28. | Day 28 after the study vaccination
GMT of neutralizing antibodies to Delta (B.1.617.2) variant on D90 and D180. | Day 90 and Day 180 after the study vaccination
GMT of neutralizing antibodies to Omicron (B.1.1.529) variant on D90 and D180. | Day 90 and Day 180 after the study vaccination
Incidence and severity of solicited AEs from D0 to D7 after study vaccination. | Day 0 to Day 7 after the study vaccination
Incidence and severity of unsolicited AEs from D0 to D28 after study vaccination. | Day 0 to Day 28 after the study vaccination
Incidence and severity of SAEs and AESIs within 180 days after study vaccination. | Day 0 to Day 180 after the study vaccination
GMT of neutralizing antibodies against SARS-CoV-2 variants other than Delta and Omicron variants on D28. | Day 28 after the study vaccination